CLINICAL TRIAL: NCT03849677
Title: Differential Analysis of Uric Acid Metabolism, Endothelial Function, Oxidative Stress and Cardiovascular Parameters in Vegans and Omnivores.
Brief Title: Uric Acid Metabolism, Endothelial Function and Oxidative Stress in Vegans and Omnivores.
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other); Fonds Erasme (Unknown); Fonds pour la chirurgie cardiaque (Unknown)
Responsible Party: Sponsor
Other Study IDs: 34735921
Record Dates: First submitted 2019-02-06; First posted 2019-02-21 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Healthy; Diet Modification
Keywords: uric acid; hemodynamic parameters; endothelial function; oxidative stress and inflammation; vegan; omnivore
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Omnivore
  Interventions: Other: Endothelial function and inflammation
- Vegan
  Interventions: Other: Endothelial function and inflammation

INTERVENTIONS:
Other: Endothelial function and inflammation — Analysis of endothelial function, oxidative stress

SUMMARY:
50 vegans and 50 omnivores will be recruited at the Erasme Hospital, Brussels.

Hypothesis

* Relative induced-hyperuricemia by the vegan diet is not associated with impaired endothelial function if vitamin B12 and folic acid levels are normal.
* Quantification of xanthine oxidoreductase (XOR) isoforms varies according to the diet. Omnivores present more xanthine oxidase (XO) than vegans in which the xanthine dehydrogenase (XD) isoform is more prevalent.
* The vegan group has more favorable oxidant, metabolic and inflammatory profiles than the omnivore group.

DETAILED DESCRIPTION:
Non-meat eaters rise widely worldwide. This choice answers ideological, ecological or health concerns. Several vegetarian diets exist and the vegan diet is the most restricted one as it excludes all animal products, eggs and dairy.

Beside benefits on health and particularly on the cardiovascular system (blood pressure, weight, lipid profile), some authors described less favorable lipid and oxidative profiles and others described an impairment in endothelial function markers in 'vegans'. These effects were attributed to low vitamin B12 and folate levels and high homocystein levels. However, vitamin B12 supplementation improved these parameters. Epidemiological studies also showed that 'vegans' disclose higher uric acid levels than other vegetarians or omnivores. Uric acid acts as an antioxidant in the plasma but can be deleterious for vascular cells leading to endothelial dysfunction. The main enzyme involved in uric acid metabolism is xanthine oxidoreductase which exists under two interconvertible isoforms. Xanthine dehydrogenase is the main form and uses nicotinamide adenine dinucleotide (NAD+) as electron acceptor and does not produce reactive oxygen species (ROS). In contrast, the other isoform xanthine oxidase uses oxygen as an electron acceptor and produces reactive oxygen species (ROS). The investigators wish to test the hypothesis that it is not uric acid per se, but which isoform of xanthine oxidoreductase which alters endothelial function. This is why the investigators wish to determine if regular 'vegans' (with normal vitamin B12 and folate levels) disclose increased uric acid levels in the presence of a reduced inflammation, oxidative stress and improved endothelial function, as compared to matched 'omnivores'.

50 vegans and 50 omnivores will be recruited at the Erasme Hospital, Brussels.

Hypothesis

* Relative induced-hyperuricemia by the vegan diet is not associated with impaired endothelial function if vitamin B12 and folic acid levels are normal.
* Quantification of oxidoreductase (XOR) isoforms varies according to the diet. Omnivores present more xanthine oxidase (XO) than vegans in which the xanthine dehydrogenase (XD) isoform is more prevalent.
* The vegan group has more favorable oxidant, metabolic and inflammatory profiles than the omnivore group.

ELIGIBILITY:
Inclusion Criteria:

* Vegan or omnivore diet for at least one year (matched for age, gender, BMI, socio-economic status and weight)
* Healthy

Exclusion Criteria:

* Smoking
* Chronic treatment
* No allowed drugs taking
* Excessive alcohol consumption

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited upon invitation on social network mainly.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Measure of the perfusion of the microcirculation of the skin | 2 hours
  Endothelial function assessment will be performed through analyse of the perfusion of the microcirculation of the skin in the forearm will be assessed by means of a laser Doppler imager and iontophoresis of acetylcholine and sodium nipride. Heating-induced hyperemia will be assessed after iontophoresis of inhibitor of NO synthase and saline. Units are perfusion unit.
  Iontophoresis is a non-invasive tool which permits to infuse molecules in the first micrometers of the skin. The used molecules are vasodilative, saline or NO synthase inhibitor.

SECONDARY OUTCOMES:
Concentration of Uric acid | 2 hours
  Uric acid (mg/dL or SI)
Concentration of xanthine oxidase and xanthine dehydrogenase in blood | 2 hours
  western blot
Measure of hemoglobin | 2 hours
  g/l
Measure of white blood cells, red blood cells and platelets | 2 hours
  cells/µl of blood
Measure of urea, creatinine, bilirubin, albumine, prealbumin, LDL, HDL, lp(a), total cholesterol, triglyceride, apolipoprotein A and B | 2 hours
  mg/dl
Measure of glycemia, vitamine and iron status (B3, B6, B12, C, D, E, B9, Zn, Cu, Selenium, iron, ferritin), c-reactive protein, homocystein | 2 hours
  mg/dl
Measure of sodium, potassium, chlore, phosphor, calcium, magnesium, HbA1c, omega 3 et 6 | 2 hours
  mmol/l
Measure of glomerular filtration rate | 2 hours
  ml/min
Measure of gamma-glutamyltransferase, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, creatin phosphokinase, insulin, TSH | 2 hours
  u/l
Measure of allantoin, homocitrulline/lysine, chloro-tyrosine/tyrosine, Il-8, myeloperoxidase | 2 hours
  Mass spectrometry and Elisa Kits
Measure of renin, aldosterone, angiotensin 2, angiotensin converting enzyme | 2 hours
Measure of main proteomes and metabolomes in cells incubated with sera from participants | 2 hours
  Sera will be used for cell cultures. Theses cells will be lysed and used to analyse and compare the different proteomes / metabolomes according to the groups. We will be able to understand which protein groups are reduced or enhanced according to the diet.
Measure of blood pressure | 2 hours
  Systolic and diastolic blood pressure
Measure of baroreflex sensitivity | 2 hours
  finometer
Measure of heart rate | 2 hours
  finometer
Measure of augmentation index | 2 hours
  Assessment of the arterial stiffness
Measure of pulse wave velocity | 2 hours
  Assessment of the arterial stiffness
Diet questionary | 2 hours
  Diet History Questionnaire third version provides estimation of one year consumption of proteins, carbohydrates, lipids, micronutrient and vitamines

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme Hospital, Brussels, Belgique, Belgium

IPD SHARING:
Plan to Share IPD: No